CLINICAL TRIAL: NCT07239167
Title: A Prospective Cohort Study on Patient With Obesity Undergoing Weight Change
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202504134RINA
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Obesity & Overweight; Weight Loss; Metabolic Syndrome; Metabolic Dysfunction-Associated Steatohepatitis; Obesity (Disorder)
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- A prospective cohort study on patients with obesity undergoing weight change

SUMMARY:
This prospective cohort study collected baseline data and followed up obese patients at their first visit to a weight loss clinic. The study examined the impact of various predictors and biomarkers on weight loss outcomes, aiming to establish an evidence-based foundation for personalized weight loss treatment.

Participants underwent a battery of measurements and questionnaires, including height, weight, waist circumference, blood pressure, blood tests, and questionnaires addressing diet, exercise, stress, sleep, and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older, regardless of gender.
2. Body mass index (BMI) ≥ 27 kg/m², or ≥ 24 kg/m² with one or more obesity-related comorbidities.
3. Willing to undergo any form of weight loss intervention.
4. Able to read and understand Chinese, willing to complete questionnaires, blood tests, and follow-up follow-up.
5. Voluntarily consent to participate and be willing to complete the subject consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Individuals with significant mental illness (e.g., schizophrenia, severe depression) or cognitive impairment that may affect their ability to consent or cooperate with the study.
3. Individuals with severe organ dysfunction (e.g., end-stage renal disease, cirrhosis, congestive heart failure, etc.).
4. Individuals taking medications that significantly affect their weight (e.g., long-term steroids or antipsychotics) and cannot be discontinued.
5. Individuals deemed unsuitable for participation in this study by the study leader (e.g., individuals who are expected to be unable to complete follow-up).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participate were first diagnosed at the weight loss clinic at the National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2035-05-05 (Estimated)

PRIMARY OUTCOMES:
Baseline data were collected and followed up during the subjects' initial visit to the weight loss clinic to establish an evidence-based basis for personalized weight reduction treatment. | Weight changes of subjects after 24 weeks, 48 weeks, 72 weeks, and 96 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- No.7, Chung Shan S. Rd.（Zhongshan S. Rd.）, Taipei, Zhongzheng Dist, Taiwan